CLINICAL TRIAL: NCT03805139
Title: Role of Ajwa Derived Polyphenols in Dyslipidaemias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, NASEER AHMED, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Dyslipidemias; Hyperglycemia; Liver Dysfunction; Oxidative Stress; Hemoglobin SC; Anemia
Keywords: Ajwa (Pheonix Dactylfera) Derived polyphenol; Dyslipidemia; Cardioprotection; HDL; Transferulic Acid; Gallic Acid
MeSH Terms: conditions — Dyslipidemias; Hyperglycemia; Liver Diseases; Hemoglobin SC Disease; Anemia

STUDY DESIGN:
Intervention Model Description: A total of 60 subjects (30 in each group) will be included in the study. The total duration of study will be upto 6 months. The AKU faculty and staff will be invited to MDL lab for screening and initial baseline, enrolled participant will be informed for inclusion in the research on the basis of our criteria of HDL levels. Written informed consent (a copy will also be provided to the participant) will be taken from each individual. A questionnaire regarding their diet and life style will be filled. Following vitals will be measured body weight, height and blood pressure. Blood sample will be taken for lipid profile (LDL, HDL, total cholesterol and triglycerides). Total period for each participant will be 6 weeks for interventions. In Ajwa Dates group, number of interaction will be 5 days a week for 6 weeks (30 doses will be provided).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ajwa Dates group (Experimental): 55-65gms Ajwa dates 7 days a week for 6 weeks
  Interventions: Dietary Supplement: Ajwa Date (phoenix dactylifera)
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Ajwa Date (phoenix dactylifera) — Effect of Ajwa on Dyslipidemia
  Arms: Ajwa Dates group

SUMMARY:
World Health Organization report notifies of the escalating global burden of cardiovascular diseases (CVD), projecting that it will become the major worldwide cause of death and disability by 2020. The South Asian countries have the highest rates of CVD globally. It is widely acknowledged that South Asians have 40-60% higher risk of CVD linked to mortality, compared with other populations. Multiple human population studies have established the concentration of high density lipoprotein (HDL) cholesterol as an independent, inverse predictor of the risk of having a cardiovascular event. Furthermore, HDLs have several well-documented functions with the potential to protect against cardiovascular disease. This study trial is designed to find out the role of alternative medicine such as functional food to improve the dyslipidemia and particularly increase the levels of HDL in general population. We expect that the use of Ajwa dates will significantly enhance the level of HDL and reduce cardiovascular events in general population.

DETAILED DESCRIPTION:
Overall lipid profile is important in cardiovascular diseases but particularly serum HDL levels have long been recognized as an independent inverse prognostic marker of CVD, when the Framigham study, in 1980s showed that HDL below 40-60mg/dl is of prognostic relevance. A rise of 1mg/dl in HDL levels is considered to reduce coronary artery disease (CAD) risk to 2-3%. Even patients with elevated total cholesterol (TC) and LDL, presenting a high HDL are seen to be protected from atherosclerosis. Multiple human population studies have shown the concentration of HDL cholesterol as an independent, inverse predictor of the risk of having a cardiovascular event. Additionally, HDL has several well-documented functions with the potential to protect against cardiovascular diseases. These include an ability to promote the efflux of cholesterol from macrophages in the artery wall, inhibit the oxidative modification of LDL, inhibit vascular inflammation, inhibit thrombosis, promote endothelial repair, promote angiogenesis, anti-oxidant, enhance endothelial function, improve diabetic control, and inhibit hematopoietic stem cell proliferation. HDL also exerts direct cardio protective effect, which are mediated with its interactions with the myocardium.

Various studies have emphasised the high incidence of CVD within the South Asian countries. The increased risk of cardiovascular events in South Asians at a younger age might be due to unknown factors affecting plaque rupture, the interaction between prothrombotic factors and atherosclerosis, or may be due to any undiscovered risk factors. Urbanisation and westernisation is characterised by a distinct increase in the intake of energy dense foods, a decrease in physical activity, and a heightened level of psychosocial stress, all of which promote the development of hyperglycaemia, hypertension, and dyslipidaemia. Most common dyslipidaemia in South Asians is low HDL-C and high triglycerides. High triglyceride and low HDL-C levels are metabolically interlinked. This metabolic phenotype is also associated with increased levels of small LDL particles despite relatively normal levels of LDL-C among South Asians. This clinical syndrome is accompanied by insulin resistance, a condition frequently referred to as atherogenic dyslipidemia, which is a common metabolic derangement among Asian. South Asians not only have lower HDL levels but also have a higher concentration of small, less-protective HDL particles. One proposed mechanism is presence of dysfunctional HDL particles. Another potential explanation for the apparent blunted cardioprotection of HDL in South Asians might be related to HDL particle size. Small particles might be less efficient in reverse cholesterol transport. In general, HDL particle size tends to be lower in patients with CHD and those with low HDL-C levels . Alarmingly, an estimated 60-80% of Pakistani population has been reported to have low HDL. There are a number of non-pharmacological and pharmacological recommendations for management of low HDL. Non-pharmacological (functional food) strategies are reported to increase HDL levels around 10-15% and which include regular exercise , body weight reduction in obese individuals , cessation of cigarette smoking in smokers and dietary modifications like decrease intake of saturated trans-fatty acids with increase intake of omega-3 polyunsaturated fatty acids . There are also a number of pharmacological agents being considered as therapeutic options but the tolerability and safety issues limit their use in addition to limited success in improving HDL. Therefore, the focus of research now days had been toward the use of functional food which can play significant role in cardiac protection. Ajwa dates have been recognized to contain the nutritional and medicinal properties. These are a rich source of nutrition, containing sugars, proteins, vitamins, high dietary fibres, minerals and fats, various phytochemicals like sterols, polyphenols, flavonoids and glycosides. Ajwa fruit is gifted by nature and is enriched with polyphenols and can act as a protective agent against many diseases. Various studies have been conducted to investigate the presence of different polyphenols in Ajwa. Different researchers have determined different phenolic components

ELIGIBILITY:
INCLUSION CRITERIA:

* General population from AKU with serum HDL < 40 mg/dl for men and women
* Adult ages (18- 70years ) will be included in the study.

EXCLUSION CRITERIA:

* Individuals with Dates/Ajwa allergy
* Individuals Patients already taking regular Ajwa
* Pregnant women and individuals with diabetes, metabolic syndrome or any other co-morbidity will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-12-07 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | 6 weeks
  Increase in HDL 3mg/dl, decrease LDL, TG, TC reduction in LDL, Triglycerides, total cholesterol 5mg/dl
Lipid profile | 6 weeks
  reduction in LDL
Lipid profile | 6 weeks
  reduction in triglycerides
Lipid profile | 6 weeks
  reduction in Total cholesterol
Lipid profile | 6 weeks
  Increase in HDL 3mg/dl reduction in LDL, Triglycerides, total cholesterol 5mg/dl
Lipid profile | 6 weeks
  reduced insulin resistance reduction in LDL, Triglycerides, total cholesterol 5mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1.Rocha-Guzmán NE, Herzog A, González-Laredo RF, Ibarra-Pérez FJ, Zambrano-Galván G, Gallegos-Infante JA: Antioxidant and antimutagenic activity of phenolic compounds in three different colour groups of common bean cultivars (Phaseolus vulgaris). Food Chemistry 2007, 103:521-527. 2. Majewska-Wierzbicka M, Czeczot H: [Flavonoids in the prevention and treatment of cardiovascular diseases]. Polski merkuriusz lekarski : organ Polskiego Towarzystwa Lekarskiego 2012, 32:50-54. 3. Salvamani S, Gunasekaran B, Shaharuddin NA, Ahmad SA, Shukor MY: Antiartherosclerotic effects of plant flavonoids. BioMed research international 2014, 2014:480258. 4. Norata GD, Marchesi P, Passamonti S, Pirillo A, Violi F, Catapano AL: Anti-inflammatory and anti-atherogenic effects of cathechin, caffeic acid and trans-resveratrol in apolipoprotein E deficient mice. Atherosclerosis 2007, 191:265-271. 5. Riccioni G, Gammone MA, Tettamanti G, Bergante S, Pluchinotta FR, D'Orazio N: Resveratrol and anti-atherogenic effects. International journal of food sciences and nutrition 2015, 66:603-610.